CLINICAL TRIAL: NCT06860204
Title: Cutting Weight, Gaining Stress: the Hidden Battle That Outweighs Fight Day Tension in Kickboxing
Brief Title: Weight Cut Stress: the Hidden Struggle Beyond Fight Day
Status: Completed | Type: Observational
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Salih ÇABUK, Res. Ass. (Researcher), Erzurum Technical University
Other Study IDs: ETU-REC-2024-10
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HRV; Psychological Adaptation
Keywords: Rapid weight loss; weight-cutting; elite kickboxers; heart rate variability; RMSSD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- weight-cutting group: Athletes in the weight-cutting group were defined as those who had lost at least 5% of their body weight within the 48 hours prior to weigh-in.
- control group: Participants in the non-weight-cutting group did not engage in any weight-cutting procedures

SUMMARY:
This study investigated the effects of rapid weight-cutting on stress in elite kickboxers by analyzing Heart Rate Variability (HRV) and subjective stress levels using a Visual Analog Scale (VAS). Data were collected across seven time points: Weigh-in Morning, Pre-Weigh-in, Post-Weigh-in, Post-Weigh-in Meal, Match Day Morning, Pre-Match, and Post-Match. Participants were divided into a weight-cutting group (n = 12), who reduced at least 5% of their body weight within 48 hours before competition, and a control group (n = 13), who maintained regular training and nutrition. HRV was measured using Apple Watch photoplethysmography under real-world conditions during the Senior European Kickboxing Championship in Greece. Results showed consistently lower RMSSD, indicating sustained physiological stress in the weight-cutting group. Subjective stress levels were also higher in this group, peaking before the weigh-in and exceeding pre-match levels. A notable decrease in subjective stress was observed immediately after the weigh-in, attributed to psychological relief rather than physical recovery. However, low RMSSD persisted on match day, indicating incomplete physiological recovery despite stabilized subjective stress. The control group demonstrated stable HRV and VAS. These findings highlight the prolonged autonomic strain of rapid weight-cutting, emphasizing the need for careful management to safeguard athlete health and performance.

DETAILED DESCRIPTION:
Objective:

This study aims to investigate the effects of rapid weight-cutting on objective (Heart Rate Variability - HRV, measured via RMSSD) and subjective (Visual Analog Scale - VAS) stress parameters in elite kickboxers. The evaluation will occur across seven specific time points: Weigh-in Morning, Pre-Weigh-in, Post-Weigh-in, Post-Weigh-in Meal, Match Day Morning, Pre-Match, and Post-Match.

Study Design:

An observational comparative design will be employed to assess objective and subjective stress responses related to weight-cutting in elite kickboxers. The study will take place during the Senior European Kickboxing Championship in Greece, from November 2 to November 10, 2024, under real competition conditions. Two groups will be included: a weight-cutting group and a non-weight-cutting group. This design will enable comparisons between objective (RMSSD) and subjective (VAS) stress measures, as well as between athletes who reduce weight and those who do not. Data will be collected at seven key time points to capture stress variations during the weight-cutting and competition phases.

Participants:

Elite kickboxers will be selected based on specific inclusion criteria. A sample size calculation using G*Power, based on an ANOVA with repeated measures and within-between interaction, determined a minimum of 22 participants to ensure adequate statistical power. Parameters include an effect size of 0.25, an alpha level of 0.05, and a power of 0.90. Accounting for potential data loss, the study targets 25 participants, with 12 in the weight-cutting group and 13 in the non-weight-cutting group. Participants will be active male elite kickboxers, aged 18-35, with at least five years of national or international competitive experience. The weight-cutting group will consist of athletes losing at least 5% of their body weight within 48 hours before the weigh-in, while the non-weight-cutting group will include those with no weight-cutting procedures and a maximum weight loss of 2% during pre-weigh-in training. Participation will be voluntary, with athletes provided detailed information about the study's purpose, methods, and risks, and written informed consent will be obtained. Confidentiality will be ensured, and data will be used solely for research purposes. The study has been approved by the Erzurum Technical University Scientific Research and Publication Ethics Committee (Meeting No: 10, Decision No: 10, Date: 12.09.2024).

Data Collection:

Data collection will focus on objective and subjective stress parameters using HRV and VAS. Objective stress will be measured via RMSSD values, recorded with Apple Watch Series 8 devices equipped with photoplethysmography technology. Participants will wear the device in a calm, seated position for five-minute intervals to ensure reliable HRV data. Subjective stress will be assessed using the VAS, where participants rate their perceived stress on a scale. Measurements will occur at seven time points surrounding the weigh-in and competition period: Weigh-in Morning, Pre-Weigh-in, Post-Weigh-in, Post-Weigh-in Meal, Match Day Morning, Pre-Match, and Post-Match.

Data Analysis:

Data will be analyzed using SPSS version 26. Pairwise group comparisons will use Hedges' g effect size calculations, adjusted for small sample sizes, and interpreted classification (trivial < 0.2, small 0.2-0.59, moderate 0.60-1.19, large 1.20-1.99, very large 2.0-3.99, nearly perfect > 4.0). Changes across the seven time points for RMSSD and VAS will be examined with repeated measures ANOVA, including within-between interactions. Significant effects or interactions will be followed by Bonferroni-adjusted post hoc tests to control for multiple comparisons. Partial eta-squared (η²ₚ) values will be reported to evaluate practical significance. Statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Elite male kickboxers aged between 18 and 35 years
2. Minimum 5 years of competitive experience at the national or international level
3. Actively competing in the Senior European Kickboxing Championship
4. For the weight-cutting group: Must have lost at least 5% of body weight within the 48 hours prior to weigh-in

Exclusion Criteria:

1. Athletes who lost between 3-4% of their body weight, as they do not fit into either group
2. History of cardiovascular diseases
3. History of metabolic disorders
4. Any medical condition that could affect HRV measurements
5. Current or recent injuries (within the last 3 months) that could impair performance or stress responses

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consisted of elite male kickboxers competing at the Senior European Kickboxing Championship in Greece. Participants were aged 18 to 35 years and had a minimum of 5 years of competitive experience at the national or international level.
  Athletes were divided into two groups:
  Weight-Cutting Group (n = 12): Athletes who lost at least 5% of their body weight within 48 hours prior to weigh-in.
  Control Group (n = 13): Athletes who maintained their regular training and nutrition, with no more than 2% weight fluctuation before the competition.
  All participants underwent heart rate variability (HRV) assessments using photoplethysmography (PPG) via Apple Watch Series 8 and subjective stress evaluations using the Visual Analog Scale (VAS) at seven time points from weigh-in morning to post-match.
  Participants were selected based on strict inclusion and exclusion criteria to ensure comparability between groups.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) - RMSSD Changes Over Time | Baseline (Weigh-in Morning), immediately before weigh-in, immediately after weigh-in, post-weigh-in meal, morning of match day, immediately before match, immediately after match
  Heart Rate Variability (HRV) was assessed using the Root Mean Square of the Successive Differences (RMSSD) to evaluate autonomic nervous system stress responses. RMSSD values were measured to determine the impact of rapid weight-cutting on physiological stress and recovery. Lower RMSSD values indicate higher physiological stress and impaired autonomic function.

SECONDARY OUTCOMES:
Subjective Stress Levels (VAS Scores) Over Time | Baseline (Weigh-in Morning), immediately before weigh-in, immediately after weigh-in, post-weigh-in meal, morning of match day, immediately before match, immediately after match
  Subjective stress levels were assessed using the Visual Analog Scale (VAS), where participants rated their perceived stress from 0 (no stress) to 10 (extreme stress). Measurements were taken to evaluate the psychological impact of rapid weight-cutting. Higher VAS scores indicate greater subjective stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Faculty of Sport Sciences, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with researchers upon reasonable request. The following data will be available:
  Heart Rate Variability (HRV) data (RMSSD values) collected at seven time points Visual Analog Scale (VAS) stress scores at seven time points Basic demographic data (age, weight category, competition level)
  Access and Conditions:
  Data will be available after study publication for researchers conducting related studies in sports science, physiology, or psychology.
  Researchers must submit a formal request, including a study proposal, to the corresponding author (Burak Karababa, burak.karababa@erzurum.edu.tr).
  Access will be granted upon approval and agreement to data use terms, ensuring confidentiality and ethical research practices.
Supporting Information: SAP, Analytic Code
Time Frame: Start Date: Data will be available upon publication of study results (estimated [insert expected publication year, e.g., 2025]).
  End Date: Data will be available for 5 years after publication or until [insert expected end year, e.g., 2030], whichever comes first.
Access Criteria: Researchers affiliated with academic institutions, sports science organizations, or health research centers conducting studies related to sports physiology, combat sports, weight-cutting, stress, or heart rate variability (HRV).
  Access will be granted only to those with a valid research proposal that aligns with the objectives of this study.
  Researchers must submit a formal request, including a study proposal and intended data use statement, to the corresponding author (Burak Karababa, burak.karababa@erzurum.edu.tr).
  Upon approval, data will be shared via secure data transfer methods (e.g., institutional repository, encrypted file sharing platform).
  Researchers must agree to data use terms, including confidentiality and ethical compliance, before accessing the dataset.